CLINICAL TRIAL: NCT02858843
Title: A Study of the Effect of Combination Lumacaftor and Ivacaftor on Markers of Hyperglycemia in Persons With Cystic Fibrosis
Brief Title: The Effect of Combination Lumacaftor and Ivacaftor on Markers of Hyperglycemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to enroll eligible subjects for the study.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jose C. Florez, MD, PhD, Chief of the Diabetes Unit, Associate Professor Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2016P000959
Record Dates: First submitted 2016-07-05; First posted 2016-08-08 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Cystic Fibrosis; Diabetes
Keywords: genetics
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lumacaftor-ivacaftor (Experimental): Subjects will be monitored for glycemic changes before and after starting lumacaftor-ivacaftor.
  Interventions: Drug: lumacaftor-ivacaftor

INTERVENTIONS:
Drug: lumacaftor-ivacaftor — Drug given for cystic fibrosis
  Other Names: Orkambi

SUMMARY:
The purpose of this research study is to find out if the combined therapy lumacaftor-ivacaftor affects glycemia in patient with cystic fibrosis.

DETAILED DESCRIPTION:
This is a single center, open label study. Patients will have 1 visits at the Diabetes Research Center (DRC), or Clinical Research Center (CRC).

The participants will have been previously screened to make sure they are candidates for the study. These patients will be contacted prior to their first visit to discuss enrollment in the study.

At the study visit the participant will come to the CRC or DRC for a research visit. The following will occur at this study visit: informed consent; brief medical history; weight and height; vital signs and blood pressure; blood draw for DNA extraction, A1c and an extra research tube for storage. This will be scheduled at a time that is convenient to the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old or greater
2. Patients diagnosed with cystic fibrosis (CF), genotype homozygous Phe508del
3. Subject has been started on lumacaftor-ivacaftor for clinical reasons, with no contraindication for starting the drug* * Contraindications for taking drug include abnormal liver enzyme tests, renal dysfunction, pregnancy or nursing mothers

Exclusion Criteria

1. Does not have a HgbA1c within 1 year prior to starting medication.
2. Has not been on the combination therapy for at least 2 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-08-01; Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Change in glycated hemoglobin (hemoglobin A1C) | 1 year
  A blood test will be used to determine the hemoglobin A1c change while on the medication.
Change in units of insulin used over a period of 6 months to 1 year. | 1 year
  Using chart review, the change in insulin units used per day will be calculated

SECONDARY OUTCOMES:
Change in glycemia contingent on genetic risk score | 1 year
  The investigators will examine how change in glycemia is dependent on genotype at variants associated with type 2 diabetes and insulin secretion using genetic risk scores.
Pulmonary function test (PFT) forced expiratory volume at one second (FEV1) measurements | 1 year
  The investigators will compare how PFT measurement of FEV1 are related to changes in glycemia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wainwright CE, Elborn JS, Ramsey BW, Marigowda G, Huang X, Cipolli M, Colombo C, Davies JC, De Boeck K, Flume PA, Konstan MW, McColley SA, McCoy K, McKone EF, Munck A, Ratjen F, Rowe SM, Waltz D, Boyle MP; TRAFFIC Study Group; TRANSPORT Study Group. Lumacaftor-Ivacaftor in Patients with Cystic Fibrosis Homozygous for Phe508del CFTR. N Engl J Med. 2015 Jul 16;373(3):220-31. doi: 10.1056/NEJMoa1409547. Epub 2015 May 17. PMID 25981758
- [Background] Bellin MD, Laguna T, Leschyshyn J, Regelmann W, Dunitz J, Billings J, Moran A. Insulin secretion improves in cystic fibrosis following ivacaftor correction of CFTR: a small pilot study. Pediatr Diabetes. 2013 Sep;14(6):417-21. doi: 10.1111/pedi.12026. Epub 2013 Mar 13. PMID 23952705